CLINICAL TRIAL: NCT06572423
Title: Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy for Palliative Head and Neck Cancer Treatment (PULS-Pal)
Acronym: PULS-Pal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-000663
Record Dates: First submitted 2024-08-16; First posted 2024-08-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Carcinoma; Localized Head and Neck Carcinoma; Metastatic Head and Neck Carcinoma; Recurrent Head and Neck Carcinoma
MeSH Terms: interventions — DEAE-Dextran; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; X-Rays; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (PULSAR and HyperArc) (Experimental): Patients undergo standard of care CT simulation for radiation treatment planning using HyperArc software. 1 week later, patients undergo PULSAR fraction therapy once daily on days 0, 14, 28, 42, and 56. Patients may also undergo Positron Emission Tomography (PET) scan and MRI during follow-up.
  Interventions: Procedure: Personalized ultrafractionated stereotactic adaptive radiotherapy; Radiation: Volume Modulated Arc Therapy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Other: Best Practice; Behavioral: University of Washington Quality of Life Scale, Version 4; Behavioral: Functional Assessment of Cancer Therapy-Head & Neck

INTERVENTIONS:
Procedure: Personalized ultrafractionated stereotactic adaptive radiotherapy — PULSAR is a radiation therapy regimen that uses a limited number of fairly large dose pulses while adjusting to specific anatomic and/or biological changes which may occur during the course of the treatment.
  Other Names: PULSAR
Radiation: Volume Modulated Arc Therapy — Use HyperArc technology
  Other Names: VMAT; Volumetric Modulated Arc Therapy
Procedure: Computed Tomography — Undergo CT simulation for radiation planning
  Other Names: CAT; CAT Scan; Computed Axial Tomography; CT; CT Scan
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging; PET; PET Scan; proton magnetic resonance spectroscopic imaging
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; MRI
Other: Best Practice — Undergo standard of care
  Other Names: standard of care
Behavioral: University of Washington Quality of Life Scale, Version 4 — Complete questionnaire
  Other Names: UW QOL v4
Behavioral: Functional Assessment of Cancer Therapy-Head & Neck — Complete questionnaire
  Other Names: FACT Head and Neck Questionnaire; FACT-H&N Questionnaire

SUMMARY:
This trial tests how well personalized ultra fractionated stereotactic adaptive radiotherapy (PULSAR) works together with HyperArc© radiation treatment planning technology for palliative (holistic pain and symptom control) tumor control in patients with primary or recurrent, localized or metastatic head and neck cancer (HNC) who are ineligible for or decline standard of care treatment. Researchers want to evaluate if using HyperArc and PULSAR together will deliver higher, possibly more effective doses, resulting in better tumor control with the same or fewer side effects than smaller routine doses. PULSAR is a radiation therapy regimen that uses a limited number of fairly large dose pulses while adjusting to specific anatomic and/or biological changes which may occur during the course of the treatment. HyperArc radiation treatment planning technology is a tool that allows for target dose escalation to tumor tissue while maintaining minimal head and neck organs-at-risk doses compared to other radiation treatment planning software. Undergoing PULSAR and HyperArc technology together may be a safe and effective palliative treatment option for patients with HNC.

DETAILED DESCRIPTION:
A significant proportion of patients with de novo or recurrent head and neck cancer are not candidates for standard-of-care definitive treatment(s), including standard-of-care stereotactic body radiation therapy (SBRT). Current palliative radiation therapy regimens result in adequate symptom improvement though with suboptimal local control and/or toxicity. The durability of symptom and local control in these patients is becoming more important as advances in systemic therapy are improving these patients' survival.

After confirmation of eligibility, enrolled patients will undergo radiation simulation and planning per standard of care. HyperArc technology will be used for treatment planning given prior internal validation of its superiority. Dosimetric constraints will be adapted from the available literature as appropriate. Patients will receive an 11 Gray fraction of radiation to the head and neck tumor site every 14 +/-10 days.

It is possible that patients will experience anatomical and/or tumor changes during the radiation therapy course such that patient alignment for radiation therapy is no longer optimized to the original CT simulation and radiation plan. In such cases where it is determined that adaptive planning is needed, the Investigators will abort planned radiation therapy and immediately perform re-simulation and re-planning if the anatomic change is significant enough to put adjacent normal tissue at significant risk; otherwise, the Investigators will re-plan with the next fraction of radiation to minimize treatment delays. This will be determined by the treating physician through standard of care clinical criteria and procedures.

The frequency of re-simulation and adaptive planning as well as associated changes in dosimetry will be measured. Patients will receive 5 PULSAR fractions for a total radiation dose of 55 Gray. Treatment will be terminated early in cases of intolerable treatment-related toxicity, altered clinical context, or the patient declines further treatment.

Enrolled patients are permitted to receive systemic therapy at the discretion of their medical oncologist.

Patient follow-up will be measured from the time of receipt of first PULSAR fraction to 12 months after receipt of the last PULSAR fraction.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Diagnosis of primary or recurrent, localized or metastatic (American Joint Committee on Cancer (AJCC) 8th Edition stages I-IV) head and neck cancer. In primary diagnosis cases, pathologic confirmation is required. In recurrent and/or metastatic diagnosis cases, pathologic confirmation is not required if not beneficial to the patient as standard of care, and diagnosis can be assumed based on clinical and/or radiographic evidence
* Ineligible for or declines standard of care definitive treatment(s), which will be documented in the patient's trial screening progress note in their electronic medical record by the treating physician
* Measurable disease within the head and/or neck clinically and/or on imaging studies (CT, PET, MRI) within 30 days from date of enrollment
* Patient maximum tumor(s) or tumor bed diameter must be less than 10cm
* In a woman of childbearing potential, a negative serum or urine pregnancy test within 1 week of treatment start must be documented. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for duration of study participation and for up to 4 weeks following the study treatment
* Patients with a tracheostomy and/or a percutaneous endoscopic gastrostomy tube are eligible for inclusion

Exclusion Criteria:

* Pregnant or breast-feeding
* More than 1 prior radiation treatment course directed to the treatment area over the patient's lifetime. In patients who have received 1 prior radiation treatment course directed to the treatment area, that prior radiation treatment course must have concluded at least 6 months prior to trial enrollment
* Any comorbidity or condition which would limit full compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2028-12-16 (Estimated); Study Completion 2029-12-16 (Estimated)

PRIMARY OUTCOMES:
Time to progression of the treated tumor target | From baseline up to 1 year
  Progression of the treated tumor target will be determined clinically and/or radiographically as applicable. Time to progression of the treated tumor target will be reported descriptively for each patient. One-year treated tumor target progression free survival will be estimated by the Kaplan-Meier method, descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum), and will consider the competing risk of death.

SECONDARY OUTCOMES:
Grade 3 or higher treatment-related toxicity | Within 24 months after treatment completion
  According to the Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Will be performed across the whole cohort, as well as separate analysis stratifying patients by Human Papillomavirus/p16 status.
Disease progression free survival (PFS) | From enrollment to the first objectively documented disease progression, either in or out of the treated field per radiographic and/or clinical evaluation, or death due to any cause, assessed up to 24 months
  Disease progression of any type will be determined clinically and/or radiographically as applicable. Time to disease progression will be reported descriptively for each patient. One-year disease progression free survival will be estimated by the Kaplan-Meier method, descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum), and will consider the competing risk of death.
Overall survival (OS) | From enrollment until death due to any cause, assessed up to 24 months.
  The Kaplan-Meier method will be used to summarize overall survival.
Longitudinal patient reported outcomes on the University of Washington Quality of Life (UW-QoL) Questionnaire | From baseline up to 24 months
  Represented by changes from baseline in the pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood, anxiety, intimacy, fear of cancer recurrence, overall health-related quality of life, and overall quality of life domains. Each domain ranges from 0-100 with higher scores meaning a better outcome. Changes will be analyzed with respect to whether they represent minimally important differences.
Longitudinal patient reported outcomes on the Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) Questionnaire | From baseline up to 24 months
  Represented by changes from baseline in the physical well-being, social/family well-being, emotional well-being, functional well-being domains and additional concerns. Each domain has multiple specific questions with a 5 point Likert-type scale for responses. Changes will be analyzed with respect to whether they represent minimally important differences.
Radiation therapy dosimetry | through study completion, on average of 24 months
  Will be performed on patients included in analysis sets FAS and EAS across the whole cohort, as well as separate analyses stratifying patients by Human Papillomavirus/p16 status.
Radiation therapy planning | through study completion, on average of 24 months
  Frequency of re-simulation and/or adaptive planning required with PULSAR
Incidence of adverse events (AE) | From baseline up to 24 months
  Safety analyses will be performed for patients included in analysis set Statistical Analysis Software (SAS)

CONTACTS AND LOCATIONS:
Overall Officials: Travis Courtney, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courtney PT, L Santoso M, Savjani RR, K Reddy V, Chai-Ho W, Velez Velez MA, J Wong D, Palodichuk C, Basehart TV, P O'Connell D, Cao M, Telesca D, Chin RK. A phase II study of personalized ultrafractionated stereotactic adaptive radiotherapy for palliative head and neck cancer treatment (PULS-Pal): a single-arm clinical trial protocol. BMC Cancer. 2024 Dec 21;24(1):1564. doi: 10.1186/s12885-024-13303-5. PMID 39709372